CLINICAL TRIAL: NCT04088773
Title: Biomarkers of Intestinal Fibrosis in Small Bowel Crohn's Disease
Status: Active, not recruiting | Type: Observational
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: The Leona M. and Harry B. Helmsley Charitable Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-0677
Record Dates: First submitted 2019-09-12; First posted 2019-09-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Crohn Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Aim 1 Crohn Disease participants (B2 phenotype): Crohn's Disease participants scheduled for ileal small bowel resection; No intervention; observational only; collection of blood, stool, and perform MRI; completion of Crohn's Activity Questionnaire
  Interventions: Diagnostic Test: blood biomarkers; Diagnostic Test: stool biomarkers; Diagnostic Test: MRI imaging
- Aim 2 Crohn Disease participants (B1 phenotype): Crohn's Disease participants with uncomplicated small bowel disease; No intervention; observational only; collection of blood, stool, and perform MRI; completion of Crohn's Activity Questionnaire
  Interventions: Diagnostic Test: blood biomarkers; Diagnostic Test: stool biomarkers; Diagnostic Test: MRI imaging
- Aim 2 Healthy Controls: No intervention; observational only; collection of blood, stool, and completion of Gastrointestinal Symptoms Rating Scale
  Interventions: Diagnostic Test: blood biomarkers; Diagnostic Test: stool biomarkers

INTERVENTIONS:
Diagnostic Test: blood biomarkers — biomarkers to distinguish fibrotic vs non-fibrotic CD lesions
Diagnostic Test: stool biomarkers — fecal biomarkers of inflammation, mucosal inflammation
Diagnostic Test: MRI imaging — MRI imaging to detect bowel wall fibrosis and to detect inflamed, non-fibrotic from inflamed, fibrotic bowel
  Groups: Aim 1 Crohn Disease participants (B2 phenotype); Aim 2 Crohn Disease participants (B1 phenotype)

SUMMARY:
This research study will evaluate if specific blood, stool and MRI tests can tell the difference between bowel wall inflammation without scarring and bowel wall inflammation with scarring that can cause bowel blockages requiring surgery.

DETAILED DESCRIPTION:
This multi-center study will test the accuracy of individual and combined MRI and blood-based diagnostic tools in both children and adults with small bowel CD. We will determine the accuracy of a composite tool (including its multiple individual biomarkers) for defining the relative amounts of intestinal inflammation versus scarring in patients at the time of surgery (B2 disease) and in patients at an early stage of disease prior to complications (B1 disease).

ELIGIBILITY:
Inclusion Criteria:

* Aim 1 (CD participants)

  1. Aged 8-70 years
  2. Undergoing first surgical distal (ileal) small bowel resection for structuring (B2 phenotype) Crohn's disease as determined by CTE or MRE or ileocolonoscopy
  3. English speaking
* Aim 2 (CD participants)

  1. Age 8 to 70 years
  2. Uncomplicated inflammatory small bowel CD based on clinical CTE or MRE or ileocolonoscopy performed within 6 months prior to enrollment (CD participants only)
  3. English speaking
* Aim 2 (Control participants)

  1. Age 8 to 70 years
  2. English speaking

Exclusion Criteria:

* Aim1 (CD participants)

  1. B1 or B3 (i.e., fistula, abscess, phlegmon/inflammatory mass) CD phenotype
  2. Prior small bowel surgery, including but not limited to surgical resection, stricturoplasty, or endoscopic treatment of a small bowel stricture
  3. Anything to eat or drink within 4 hours of study visit (participants may take their required medications with a little water)
  4. Known pregnancy (Note: Institutional policies/procedures will be followed for pregnancy screening)
  5. Contraindication for MRI (e.g., surgical implant, claustrophobia). Note: To be determined based on local procedures.
* Aim 2 (CD participants)

  1. Stenotic ileocecal valve at colonoscopy
  2. Prior small bowel surgery, including but not limited to surgical resection, stricturoplasty, or endoscopic treatment of a small bowel stricture
  3. Anything to eat or drink within 4 hours of study visit (participants may take their required medications with a little water)
  4. Known pregnancy (Note: Institutional policies/procedures will be followed for pregnancy screening)
  5. Contraindication for MRI (e.g., surgical implant, claustrophobia). Note: To be determined based on local procedures.
* Aim 2 (Control participants)

  1. Any known gastrointestinal tract disease
  2. Any known inflammatory/autoimmune disease involving another organ system (e.g., rheumatoid arthritis, scleroderma, multiple sclerosis).
  3. Fecal calprotectin level of ˃100 mcg.gm will be excluded from further analysis and replaced.

Ages: 8 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Aim 1 - Children and adults undergoing surgical small bowel resection for structuring CD; Aim 2 - children and adults that have known uncomplicated inflammatory small bowel CD (B1phenotype) AND healthy non-IBD participants
Sampling Method: Non-Probability Sample
Enrollment: 232 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Magnetization transfer ratio (MTR) | Day 1
  compare MTR values between Aim 1 and Aim 2 cohorts

SECONDARY OUTCOMES:
Correlation between MTR values and bowel wall collagen measurements | Day 1
  combine all subjects from Aim 1 and Aim 2 that undergo MRI

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Dillman, MD, MSc, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (4):
- United States (4):
  - Emory/Children's Healthcare of Atlanta, Atlanta, Georgia
  - Michigan Medicine, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: No